CLINICAL TRIAL: NCT00150033
Title: Development and Validation of a Thyroid-Specific Quality of Life Measure
Brief Title: Health-Related Quality of Life for Thyroid Patients
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Torquil Watt, MD, Copenhagen University Hospital Rigshospitalet
Other Study IDs: 011
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Thyroid Diseases
Keywords: thyroid disease; Quality of Life; Patient reported outcome; questionnaire; Quality of Life measurement
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

Thyroid diseases are frequent. They include both metabolic changes and gland enlargement (goitre). Previous research and clinical suspicion indicate that the life quality of many patients is reduced despite successful treatment. Research methods are, however, weak, and a well-tested, disease specific quality of life questionnaire is especially needed. Several treatment possibilities exist for each thyroid disease. For example, hypermetabolism can be treated with either medication, radioactive iodine or by surgery. No comparative studies of quality of life using the different treatment modalities exist.

Purpose:

To develop and evaluate a questionnaire to measure health-related quality of life in patients suffering from thyroid diseases.

Methods:

To ensure that all relevant aspects are included, the questionnaire will be developed on the basis of a systematic examination of the scientific literature and interviews with 13 physicians and 100 patients. The questionnaire will then be tested by 100 new patients. After revision, the questionnaire will be answered by 1000 patients with a view to scientifically investigate the measuring capacity of the questionnaire. This will be done using traditional psychology methods (psychometry) as well as modern statistical methods (structural equations for categorical data and "item response" models).

Relevance:

The above-mentioned questionnaire is necessary for clarifying whether these diseases reduce quality of life and, in the long-term, whether a difference in quality of life exists using the different treatment alternatives and whether treatment can be improved. It should also be included in quality protection studies, in the evaluation of new treatment modalities and possibly also in the treatment of the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients with benign thyroid disease.

Exclusion Criteria:

* Unable to complete questionnaire: must be able to read and write Danish

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2005-05; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torquil Watt, MD, Principal Investigator — Rigshospitalet, Denmark; Ulla Feldt-Rasmussen, MD, DMSc, Study Director — Copenhagen University Hospital at Herlev
Locations (1):
- Department of Endocrinology, Rigshospitalet, Copenhagen, Sealand, Denmark

REFERENCES:
- [Background] Watt T, Groenvold M, Rasmussen AK, Bonnema SJ, Hegedus L, Bjorner JB, Feldt-Rasmussen U. Quality of life in patients with benign thyroid disorders. A review. Eur J Endocrinol. 2006 Apr;154(4):501-10. doi: 10.1530/eje.1.02124. PMID 16556711
- [Result] Watt T, Hegedus L, Rasmussen AK, Groenvold M, Bonnema SJ, Bjorner JB, Feldt-Rasmussen U. Which domains of thyroid-related quality of life are most relevant? Patients and clinicians provide complementary perspectives. Thyroid. 2007 Jul;17(7):647-54. doi: 10.1089/thy.2007.0069. PMID 17696835